CLINICAL TRIAL: NCT03483129
Title: Examining the Feasibility of Conducting a Randomised Control Trial to Evaluate the Effectiveness of a Focused 15-minute One-to-one Consultation to Improve Blood Glucose Control in Pre-diabetes
Brief Title: 15-minute Individual Consultation to Improve Blood Glucose Control in Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aberystwyth University (Other)
Collaborators: Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 239910
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Pre-Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into either the intervention or the control group. Participants in INT will receive a 15 minute one to one consultation with a nurse at their general practice. The consultation will provide the participant with information regarding the benefits of physical activity and healthy eating. Emphasis will placed on the importance of achieving at least 150 minutes of moderate physical activity each week as well as adhering to healthy dietary habits, based on the NHS Eatwell Guide. Participants will have the opportunity to discuss pre-diabetes with a nurse and ask any questions they may have. Participants placed in CON will not receive the consultation and will only attend visits to the WARU. A subgroup of participants will also be randomised for additional physical activity monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consultation (Experimental): The consultation will provide the participant with one to one information regarding the benefits of physical activity and healthy eating. Emphasis will placed on the importance of achieving at least 150 minutes of moderate physical activity each week as well as adhering to healthy dietary habits, based on the NHS Eatwell Guide (Eatwell Guide, 2016). Furthermore, participants will have the opportunity to discuss pre-diabetes with a trained practice nurse and ask any questions they may have.
  Interventions: Behavioral: Consultation
- Control (No Intervention): All participants will receive an information leaflet detailing pre-diabetes, the associated risks and steps that can be taken to avoid developing diabetes.

INTERVENTIONS:
Behavioral: Consultation — 15 minute, one to one consultation with a trained practice nurse at a GP surgery. Participants will have the opportunity to discuss pre-diabetes, the risks of developing diabetes and the steps that can be taken to improve lifestyle behaviors and reduce the risk of diabetes development.
  Arms: Consultation

SUMMARY:
This research will assess the feasibility of conducting a randomised control trial to evaluate the effectiveness of a 15-minute one-to-one consultation to improve blood glucose control in pre-diabetes. The consultation will take the form of a 15-minute one-to-one consultation between a health-care practitioner and the patient in a primary care setting. Patients with a glycated haemoglobin (HbA1c) of between 42 and 47 mmol·mol-1 will be identified in general practise and will be eligible to participate. They will attend testing sessions at baseline (before the consultation), and at three months and six months post consultation. Body mass index (BMI), waist and hip girth, blood pressure and body composition will be recorded and blood analysed for HbA1c, cholesterol and dietary components. For a three-week period following each visit, urine will be collected, a 5-ml sample on nine occasions, and physical activity will be recorded in a sub group of participants. Urine will be analysed by flow infusion electrospray mass spectrometry (FIE-MS) to determine the metabolic content, providing an indication of the diet over the three-week sampling period. The research objectives are to assess the effectiveness of recruitment strategy and willingness of patients to engage in, and adhere to, the research process; to determine the impact of consultation on health outcome measures, including HbA1c, and to establish participant and practitioner perspectives of the consultation.

DETAILED DESCRIPTION:
Participants will be required to visit the Wellbeing Assessment Research Unit (WARU), Carywn James Building, Penglais Campus, Aberystwyth University, on 3 separate occasions, for baseline, 3 month and 6 month testing. During the baseline visit, the procedures and protocol of the study will be explained and informed consent will be received. Participant's height and body mass will be collected to calculate BMI and waist and hip girth recorded. Next, participants will be asked to sit quietly for 10 minutes in the laboratory before blood pressure is recorded from the upper non-dominant arm. Participants will remain seated prior to a 6 mL blood sample being obtained from the antecubital vein and collected into a heparinised vacutainer, with minimal stasis, using standard venepuncture methods performed by a trained member of the research team. Should patients HbA1c be outside the required values during the baseline visit, they will be informed and will take no further part in the research. WARU will inform the participant's general practicioner (GP) if their HbA1c is indicative of diabetes. Body composition will be analysed using bioelectrical impedance.

Upon completion of this phase of data collection, participants will be provided with a series of validated questionnaires to complete (to be completed at every visit unless otherwise stated). These include; the International Physical Activity Questionnaire- Short Form, Food Frequency Questionnaire (baseline and 6 months), 36-Item Short Form Survey Instrument and components of the Personal Diabetes Questionnaire (baseline). Participants will complete the questionnaires unassisted although members of the research team will be available to answer any questions the participant may have relating to the questionnaires. Lastly, participants will receive instructions on the use of the urine collection kit for dietary monitoring and the ActiGraph for physical activity monitoring (if randomised). Participants will then be free to leave the laboratory. An additional acceptability questionnaire designed by the research team will be given to participants at the end of the 6 month visit and will include questions relating to the WARU visits, 15 minute consultation (if received), urine collection and ActiGraph use. Visits will last between approximately 120 minutes and 150 minutes depending on the time taken for participants to complete the relevant questionnaires.

Following completion of the baseline visit, participants will be randomised into either the intervention group (INT) or the control group (CON). Randomisation will be achieved using a minimisation software package and will ensure that there will be only minor differences between groups in the variables used in the allocation process. Participants in INT will receive a focused 15 minute one to one consultation with a practice nurse at their registered general practice. The consultation derives from the original 30 minute protocol employed during a previous study conducted by the present research team which used 104 GP-registered patients. The first half of the 30 minute consultation in that study (led by general practice) collected baseline data (height, weight, waist circumference, blood pressure) and the second half provided patients with lifestyle advice on preventing diabetes. The consultation to be used in the proposed study does not require general practice to collect baseline data and therefore the consultation time has been reduced from 30 minute to 15 minutes. The consultation will provide the participant with one to one information regarding the benefits of physical activity and healthy eating. Emphasis will placed on the importance of achieving at least 150 minutes of moderate physical activity each week as well as adhering to healthy dietary habits, based on the National Health Service (NHS) Eat Well Guide. Furthermore, participants will have the opportunity to discuss pre-diabetes with a trained practice nurse and ask any questions they may have. Participants placed in CON will not receive the consultation and will only attend visits to the WARU. Due to logistical and financial implications, a subgroup of participants will also be randomised for additional physical activity monitoring. 5 participants from INT and 5 from CON will receive an Actigraph (see below for further information on the Actigraph).

Dietary Monitoring:

Metabolic fingerprinting and metabolic profiling of human urine is able to provide a comprehensive and quantitative snapshot of dietary exposure for 12 - 24 hrs prior to urine collection. While a single sample snapshot is not representative of an individuals' habitual dietary exposure, a series of snapshots over a prolonged time period can give a robust overview of an individual's nutritional health. Previous work has demonstrated a community based urine collection protocol as a successful and non-disruptive method for monitoring habitual diet. Participants will be provided with a urine collection kit consisting of; of non-sterile urine collection straws, additive free evacuated vacutainer tubes and a urine collection container. Once urine has been collected, the sealed vacutainer tubes will be stored in an absorbent pouch within a sealed leak-proof bag and kept in the refrigerator. All urine storage equipment and instructions are fully compliant with standards for storage of Category B biological substances. Participants will receive instructions to fill the collection container with a mid-stream urine sample (in order to minimise the possibility of bacterial contamination from urethral contaminants). Any excess urine produced which is not collected in the container should be deposited within the lavatory. The tip of the transfer straw will be submerged into the urine and a vacutainer tube inserted into the transfer straw to draw the urine into the vacutainer. Any remaining urine in the container will be deposited within the lavatory. The collection container can be rinsed with tap water after each urine sample and reused for each sample collected. Vacutainer tubes will be labelled with anonymous information including participant number, sample number, weekday/weekend sample and week number. Samples will be stored in a refrigerator at 4 degrees (ºC) for a maximum of 10 days before the samples are returned to the lab either in person or by free post for freezing at -80 ºC to await analysis. Participants will record the collection details of their urine samples onto a sample collection sheet which notes the sample number and the date and time of collection. Participants will collect 3 samples a week for 3 weeks following each WARU visit. Participants must collect two urine samples within the week on non-consecutive days (e.g. Tuesday & Thursday) and collect a third sample on either day of the weekend (Saturday/Sunday). In total, participants will collect 27 urine samples during their participation in the study. Urine samples will be analysed using laboratory based Flow Infusion High Resolution Mass Spectrometry which is an established method for dietary analysis using urine samples.

Physical Activity Monitoring:

Physical activity and sedentary lifestyle will be determined using ActiGraph following baseline, 3 months and 6 month WARU visits. Participants will be provided with written and verbal instructions on how to operate the device. Participants will choose one week within the three week urine collection period to wear the ActiGraph. Participants can choose any day within the week to begin wearing the ActiGraph but must then wear it for the following 7 days unless unfeasible to do so (e.g. swimming, bathing or showering). In this instance, participants will record at what time and the amount of time they are not wearing the ActiGraph. Should participants forget to wear the device; the same procedure will be followed. Should participants miss a whole day; they must record for an extra day directly after the 7th day. An additional sheet will be provided for participants to record any time when the device is not worn. Participants do not need to wear the ActiGraph when sleeping although they must record the time they go to sleep and at what time they wake up. Participants must fit the ActiGraph in the morning as soon as it is feasible to do so. Participants can return the ActiGraph at the end of the 7 day recording period either in person or be post.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent
* Registered with a mid-Wales GP surgery
* Glycated haemoglobin between 42 mmol·mol-1 and 47 mmol·mol-1 (< 1 year)

Exclusion Criteria:

* Under judicial control
* Unable to understand and follow instructions due to cognition or language problems
* During participant identification, general practice will exclude any patients they believe are unsuitable for study involvement, for example, terminal illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible patients recruited into the study assessed by study attendance and surgery patient records | Baseline
  Quantify the percentage (%) of patients enrolled in the study based on letters of invitation sent to eligible participants from their surgery

SECONDARY OUTCOMES:
Change in HbA1c assessed by blood Hba1c assessment | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in HbA1c (mmol)
Change in BMI assessed by aggregation of height and weight | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in BMI (kg/m2). Data on height (cm) and weight (kg) aggregated to report BMI.
Change in waist circumference assessed by anthropometric measurement | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in waist circumference (cm)
Change in hip circumference assessed by anthropometric measurement | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in hip circumference (cm)
Change in fat percentage assessed by bioelectrical impedance analysis | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in fat percentage (%)
Change in HDL assessed by blood lipid assessment | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in HDL (mmol)
Change in LDL assessed by blood lipid assessment | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in LDL (mmol)
Change in Cholesterol assessed by blood lipid assessment | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in cholesterol (mmol)
Change in physical activity level assessed by Actigraph and Physical Activity Questionnaire | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in physical activity (met minutes)
Change in the urinary concentration of metabolites of high health importance assessed by FIE-MS | Change assessed between baseline and 3 months, baseline and 6 months, 3 months and 6 months
  To determine the impact of the consultation on changes in the concentration urinary of metabolites (µM/mM) of high health importance

CONTACTS AND LOCATIONS:
Overall Officials: Rhys Thatcher, Dr, Principal Investigator — Aberystwyth University
Locations (1):
- Carwyn James Building, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be accessed by the immediate research team. Any data made available to other researchers will be anonymised and presented as mean and standard deviation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT03483129/Prot_SAP_000.pdf